CLINICAL TRIAL: NCT04912882
Title: Prognosis Predicting of CRC Patients Based on Morphology and Molecular Biomaker of Circulating Tumor Cells
Brief Title: Prognosis Predicting of CRC Patients Based on Morphology and Molecular Biomaker of CTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ZSCTC1
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Group: Training group including about 500 patients that be using to building the prognosis model
  Interventions: Diagnostic Test: Circulating tumor cell
- Validation Group: Validation group including about another 500 patients that be using to validating the prognosis model
  Interventions: Diagnostic Test: Circulating tumor cell

INTERVENTIONS:
Diagnostic Test: Circulating tumor cell — detecting circulating tumor cell pre- and post operatively

SUMMARY:
Detecting circulating tumor cells from I-IV stage colorectal cancer patients pre-and post-operatively. Analyzing the morphology and biomarkers of CTCs and builting prognosis predicting model based on the morphology and biomarkers of CTCs. Verifying the prognosis model by the survival data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;

Histologically proven colorectal carcinoma (TNM stage I-IV)

R0 resection is possible according to preoperative evaluation

Written informed consent for participation in the trial.

Exclusion Criteria:

* Primary tumor or metastases not able to be removed radically

Receiving any preoperative treatment (Including chemotherapy, radiotherapy and target therapy)

Have other malignant tumors meanwhile

Other previous malignancy within 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: I-IV stage colorectal cancer patients with resectable lesion(s) who not receive preoperative treatment
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 year
  The sensitivity of the predictive based on the number and type of circulating tumor cell
Specificity | 1 year
  The specificity of predictive model based on the number and type of circulating tumor cell

SECONDARY OUTCOMES:
AUC | 1 year
  Area under curve of the predictive model

IPD SHARING:
Plan to Share IPD: Undecided